CLINICAL TRIAL: NCT01080222
Title: A Randomized, Parallel-Group, Dose-Ranging Study to Evaluate Efficacy, Safety, Pharmacokinetics, and Antiviral Activity of VX-222 and Telaprevir in Combination With and Without Peginterferon-Alfa-2a (Pegasys®) and Ribavirin (Copegus®) in Treatment-Naïve Subjects With Genotype 1 Chronic Hepatitis C
Brief Title: A Safety and Efficacy Study of the Combination of VX-222 and Telaprevir in Treatment-Naïve Subjects With Genotype 1 Chronic Hepatitis C Virus Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study discontinued
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VX09-222-103
Record Dates: First submitted 2010-03-01; First posted 2010-03-04 (Estimated); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Chronic Hepatitis C Virus Infection
Keywords: VX-950
MeSH Terms: interventions — telaprevir; lomibuvir; Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Treatment Arm A (Experimental): Treatment Arm A was discontinued as a result of patients meeting a pre-defined stopping rule related to viral breakthrough during the first four weeks of dosing.
  Interventions: Drug: telaprevir; Drug: VX-222
- Treatment Arm B (Experimental): Treatment Arm B was discontinued as a result of patients meeting a pre-defined stopping rule relating to viral breakthrough.
  Interventions: Drug: telaprevir; Drug: VX-222
- Treatment Arm C (Experimental): * Subjects who meet pre-specified viral response criteria will stop their assigned treatment at 12 weeks.
  * Subjects who do not meet the pre-specified viral response criteria will receive peginterferon alfa-2a and ribavirin for an additional 12 weeks for a total treatment duration of 24 weeks.
  * Enrollment for this arm is complete. No additional subjects will be recruited.
  Interventions: Drug: telaprevir; Drug: VX-222; Drug: ribavirin; Biological: peginterferon-alfa-2a
- Treatment Arm D (Experimental): * Subjects who meet pre-specified viral response criteria will stop their assigned treatment at 12 weeks.
  * Subjects who do not meet the pre-specified viral response criteria will receive peginterferon alfa-2a and ribavirin for an additional 12 weeks for a total treatment duration of 24 weeks.
  * Enrollment for this arm is complete. No additional subjects will be recruited.
  Interventions: Drug: telaprevir; Drug: ribavirin; Biological: peginterferon-alfa-2a; Drug: VX-222
- Treatment Arm E (Experimental): * Subjects who meet pre-specified viral response criteria will stop their assigned treatment at 12 weeks.
  * Subjects who do not meet the pre-specified viral response criteria will receive peginterferon alfa-2a and ribavirin for an additional 24 weeks for a total treatment duration of 36 weeks.
  Interventions: Drug: telaprevir; Drug: ribavirin; Drug: VX-222
- Treatment Arm F (Experimental): * Subjects who meet pre-specified viral response criteria will stop their assigned treatment at 12 weeks.
  * Subjects who do not meet the pre-specified viral response criteria will receive peginterferon alfa-2a and ribavirin for an additional 24 weeks for a total treatment duration of 36 weeks.
  Interventions: Drug: telaprevir; Drug: ribavirin; Drug: VX-222

INTERVENTIONS:
Drug: telaprevir — tablet, 1125-mg, twice daily
Drug: VX-222 — capsule, 100-mg, twice daily
  Arms: Treatment Arm A; Treatment Arm C
Drug: ribavirin — tablet, 1000-mg for subjects weighing <75-kg or 1200-mg for subjects weighing ≥75-kg, twice daily
  Arms: Treatment Arm C; Treatment Arm D; Treatment Arm E; Treatment Arm F
Biological: peginterferon-alfa-2a — subcutaneous injection, 180-mcg, once weekly
  Arms: Treatment Arm C; Treatment Arm D
Drug: VX-222 — capsule, 400-mg, twice daily
  Arms: Treatment Arm B; Treatment Arm D; Treatment Arm E; Treatment Arm F

SUMMARY:
The purpose of this study is to assess the safety and efficacy of combination treatment with VX-222 and telaprevir administered for 12 weeks with and without peginterferon-alfa-2a and/or ribavirin. The subjects enrolled in this study are chronically infected with hepatitis C virus (HCV) genotype 1 and will not have previously received treatment for their HCV infection.

This study will include an Investigational Phase and Extension Phase. These phases will contain a Treatment Period and a Follow-up Period. All subjects will be enrolled in the Investigational Phase of this study. Subjects who fail treatment during the Investigational Phase will have the option to enter the Extension Phase at which point they will be eligible to receive peginterferon alfa-2a and ribavirin for a total of 48 weeks.

Based on an evaluation of on-treatment safety, pharmacokinetic and antiviral data from patients in each arm of the trial, Vertex may elect to enroll up to two additional treatment arms (Treatment Arm E and Treatment Arm F) that will evaluate telaprevir/VX-222-based combination therapy. The components of the treatment regimens of these arms will be selected based on clinical data that emerges from the four initially-studied regimens. If enacted, up to 25 patients are expected to enroll in each additional treatment arm.

If Treatment Arm E or Treatment Arm F is discontinued subjects meeting certain criteria will have the option to enter a telaprevir-containing Rollover Phase. Subjects who do not meet the eligibility criteria to enter the Rollover Phase may elect to enter the Extension Phase.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of non-childbearing potential
* Genotype 1 chronic hepatitis C
* Laboratory evidence of HCV infection for 6 months
* Histologic evidence of chronic hepatitis C
* Subjects who have a body mass index (BMI) of ≤35 kg/m² (BMI = weight in kg / height² in meters)
* Treatment Arm E: This arm will enroll only subjects infected with HCV genotype 1b virus
* Treatment Arm F: This arm will enroll only subjects infected with HCV genotype 1a virus

Exclusion Criteria:

* Subjects who have received any previous treatment with any approved or investigational drug or drug regimen for the treatment of hepatitis C
* Subjects with any contraindications to peginterferon alfa-2a and/or ribavirin
* Subjects with any other cause of significant liver disease in addition to hepatitis C, which may include, but is not limited to malignancy with hepatic involvement, hepatitis B, drug or alcohol-related cirrhosis, autoimmune hepatitis, hemochromatosis, Wilson's disease, nonalcoholic steatohepatitis (NASH), or primary biliary cirrhosis
* Histologic evidence of hepatic cirrhosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2010-08; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | 40 weeks
  Assessed by adverse events, physical examinations, vital signs, 12 lead electrocardiograms (ECGs), and laboratory assessments (serum chemistry, hematology, and urinalysis) vital signs, 12-lead electrocardiograms (ECGs), and laboratory assessments (clinical chemistry, hematology, and urinalysis)

SECONDARY OUTCOMES:
Proportion of Subjects Who Achieve a Sustained Viral Response | 24 weeks after the completion of the last dose of the assigned study drug treatment regimen
Undetectable HCV RNA Measurements | 36 weeks
  * Time to undetectability
  * Proportion of subjects who achieve undetectable HCV RNA levels at Week 2, Week 4, Week 8, and Week 12
  * Proportion of subjects who achieve undetectable HCV RNA levels at Week 2 and Week 8
  * Proportion of subjects who have undetectable HCV RNA levels at the end of treatment
Proportion of Subjects Who Have a Viral Breakthrough or Relapse | 60 weeks
Plasma Exposures of VX-222 and Telaprevir | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Vertex Pharmaceuticals Incorporated
Locations (21):
- United States (19):
  - La Jolla, California
  - San Francisco, California
  - Aurora, Colorado
  - Gainesville, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Lutherville, Maryland
  - Rochester, Minnesota
  - St Louis, Missouri
  - Egg Harbor, New Jersey
  - New York, New York
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Providence, Rhode Island
  - Germantown, Tennessee
  - Arlington, Texas
  - San Antonio, Texas
  - Falls Church, Virginia
- New Zealand (2):
  - Auckland
  - Christchurch

REFERENCES:
- [Derived] Jiang M, Zhang EZ, Ardzinski A, Tigges A, Davis A, Sullivan JC, Nelson M, Spanks J, Dorrian J, Nicolas O, Bartels DJ, Rao BG, Rijnbrand R, Kieffer TL. Genotypic and phenotypic analyses of hepatitis C virus variants observed in clinical studies of VX-222, a nonnucleoside NS5B polymerase inhibitor. Antimicrob Agents Chemother. 2014 Sep;58(9):5456-65. doi: 10.1128/AAC.03052-14. Epub 2014 Jun 30. PMID 24982088
- [Derived] Di Bisceglie AM, Sulkowski M, Gane E, Jacobson IM, Nelson D, DeSouza C, Alves K, George S, Kieffer T, Zhang EZ, Kauffman R, Asmal M, Koziel MJ. VX-222, a non-nucleoside NS5B polymerase inhibitor, in telaprevir-based regimens for genotype 1 hepatitis C virus infection. Eur J Gastroenterol Hepatol. 2014 Jul;26(7):761-73. doi: 10.1097/MEG.0000000000000084. PMID 24901821